CLINICAL TRIAL: NCT00352924
Title: The Main Agricultural Health Study - A Prospective Study of Cancer and Other Diseases Among Men and Women in Agriculture
Brief Title: Agriculture Health Study
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999993013; OH93-NC-N013
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Prostate Cancer; Pesticide Exposures; Lymphoma; Multiple Myeloma
Keywords: Cancer; Pesticides; Agriculture; Natural History
MeSH Terms: conditions — Prostatic Neoplasms; Lymphoma; Multiple Myeloma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of Agricultural Workers: Cohort of Agricultural Workers

SUMMARY:
The "Agricultural Health Study" (AHS) is a collaborative effort between the National Cancer Institute and the National Institute of Environmental Health Sciences. The U.S. Environmental Protection Agency and the National Institute for Occupational Safety and Health are providing support for a limited exposure assessment effort.

Initial data collection on a prospective cohort of 89,658 study subjects has been completed as of December 1997. Participants completed questionnaires that included items on pesticides used, other agricultural exposures, and work practices that modify exposure as well as on other activities that may affect either exposure or disease risks (e.g., diet, exercise, alcohol consumption, medical conditions, family history of cancer, other occupations and smoking history). Phase II of the study (1998-2003) updated information on occupational exposures, diet, work practices and medical history by means of a computer assisted telephone interview. We also collected buccal cells on sample of 34,000 study participants to assess the effect of inheritable polymorphisms and the interaction of environment and genomic predisposition.

The stimulus for this prospective investigation comes from the growing evidence that, despite a low mortality overall, farmers experience an excess of several cancers. These excesses have been observed in retrospective epidemiological studies among agricultural workers in several countries. Excess cancers are observed for the lymphatic and hematopoietic system, connective tissue, skin, brain, prostate, stomach and lips. Several of these tumors (brain, NHL, multiple myeloma, and prostate) are also increasing in the general population in many of these countries. This suggests a common set of exposures may explain the high rates in farmers and rising rates in the general population.

Farmers, their families, and other pest control workers may have contact with a variety of potentially hazardous substances including pesticides, solvents, fuels and oils, engine exhaust, dust and zoonotic viruses and other microbes. Our cohort study includes all registered pesticide applicators in Iowa and North Carolina and the spouse of applicators who are farmers. The health effects of pesticide use are the primary focus of the study. The influence of other farm exposures are also being evaluated.

The focus of the phase II follow-up period (2004-2008) is to update exposure information and health histories by means of a computer assisted interview and also following the cohort to determine disease incidence and mortality. The cohort is being followed through the cancer registries within Iowa and North Carolina, the Social Security Administration database, state vital statistics offices, National Death Index, and various in-state databases, such as the listing of registered pesticide applicators. Individuals who enrolled into the study but who are no longer at the address given during enrollment (based on subsequent attempts at follow up) have been submitted and will continue to be submitted (through NIOSH) in the standard format to the IRS under their Project 057 Taxpayer Address Request Program. Identifying data provided to the IRS include only SSN and the first four letters of last name of cohort member. IRS provides in return the most current address in IRS records if a match (SSN + all four letter of last name) is found. The purpose of this effort is to identify members of the cohort who have moved out of state, to enable adjustment of person-years for incidence and mortality calculations. Persons who have moved out of state can be followed for vital status and cause of death, but not for cancer incidence.

Continuation of the protocol will provide a valuable epidemiologic resource to help prevent cancers in the future by identifying risk factors in the rural/agricultural environment. Because more cases of important cancer outcomes occur in this cohort every year, potential cancer causes can be evaluated with increased statistical power. Larger number of cases also allows for statistical control of confounding factors, making more meaningful conclusions about cancer risk, and, for some relatively infrequent cancers, such as the lyphomas and leukemias, greater follow-up time is necessary to make any meaningful observations.

...

DETAILED DESCRIPTION:
The "Agricultural Health Study" (AHS) is a collaborative effort between the National Cancer Institute and the National Institute of Environmental Health Sciences. The U.S. Environmental Protection Agency and the National Institute for Occupational Safety and Health are providing support for a limited exposure assessment effort. Initial data collection on a prospective cohort of 89,655 study subjects has been completed as of December 1997. Participants completed questionnaires that included items on pesticides used, other agricultural exposures, and work practices that modify exposure as well as on other activities that may affect either exposure or disease risks (e.g., diet, exercise, alcohol consumption, medical conditions, family history of cancer, other occupations and smoking history). Phase II of the study (1998-2003) updated information on occupational exposures, diet, work practices and medical history by means of a computer assisted telephone interview. We also collected buccal cells on sample of 34,000 study participants to assess the effect of inheritable polymorphisms and the interaction of environment and genomic predisposition. The stimulus for this prospective investigation comes from the growing evidence that, despite a low mortality overall, farmers experience an excess of several cancers. These excesses have been observed in retrospective epidemiological studies among agricultural workers in several countries. Excess cancers are observed for the lymphatic and hematopoietic system, connective tissue, skin, brain, prostate, stomach and lips. Several of these tumors (brain, NHL, multiple myeloma, and prostate) are also increasing in the general population in many of these countries. This suggests a common set of exposures may explain the high rates in farmers and rising rates in the general population.

Farmers, their families, and other pest control workers may have contact with a variety of potentially hazardous substances including pesticides, solvents, fuels and oils, engine exhaust, dust and zoonotic viruses and other microbes. Our cohort study includes all registered pesticide applicators in Iowa and North Carolina and the spouse of applicators who are farmers. The health effects of pesticide use are the primary focus of the study. The influence of other farm exposures are also being evaluated.

ELIGIBILITY:
* INCLUSION CRITERIA:

All registered pesticide applicators in Iowa and North Carolina and the spouse and children of applicators who are farmers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective cohort of 89,655 registered pesticide applicators and spouses (57,310 applicators and 32,346 spouses of private applicators) with sufficient personal identifiers to conduct follow up activities has been assembled during the first four years of recruitment in the Agricultural Health Study, 1993-1997. The majority of applicators were asked to enroll in the AHS as they obtained or renewed their pesticide registration/licenses through the agricultural extension services of the states of North Carolina and Iowa. In the last year of enrollment, applicators who received or renewed their pesticide licenses, but were never given the opportunity to enroll due to added requirements in the testing/training class, were called and asked to complete the enrollment questionnaire over the phone. Spouses of the private applicators were also given the opportunity to enroll via the telephone.
Sampling Method: Non-Probability Sample
Enrollment: 89655 (Actual)
Dates: Start 1993-04-30

PRIMARY OUTCOMES:
Non-cancer disease incidence in pesticide applicators | Follow-up was every 5 years (to date); now to be every 3-5 years (CMS linkage)
  Evaluate non-cancer health risks associated with exposure to pesticides and other potential agricultural exposures, e.g., neurotoxicity, reproductive hazards, asthma and other respiratory diseases or symptoms, immunological toxicity, kidney disease, birth outcomes, and growth and development among offspring.
measurement of pesticide and other agricultural exposures | Follow-up was every 5 years (to date)
  Assess agricultural exposures using periodic interviews and environmental and biological monitoring
Disease risk and dietary exposures | Baseline and first follow-up only
  Identify and quantify cancer and other disease risks associated with dietary exposures and cooking practices and chemicals resulting from the cooking process.
Disease in spouses and children of farmers | Cancer as annual; now semi annual; other diseases, about 3-5 years
  Evaluate the disease risks among spouses and children of farmers that may arise from indirect contact with agricultural chemicals (e.g., ambient air drifts, pesticide residues on rugs, furniture, and other items, transferring chemicals) and nonoccupational exposures (e.g., applications to pets, in homes, and on gardens).
Cancer incidence in pesticide applicators | Was annual; now semi annually (cancer linkages)
  Identify and quantify cancer risks among men and women, whites, and minorities associated with specific direct pesticide exposures and exposures to other agricultural agents.
Agricultural exposures and biomarkers of exposure, biological effect, and biomarkers of pre-clinical disease and genetic susceptibility factors | Follow-up was every 5 years (to date); now to be every 3-5 years (CMS linkage)
  Study the relationship between agricultural exposures, the occurrence of biomarkers of exposure, biological effect, and biomarkers of pre-clinical disease and genetic susceptibility factors relevant to carcinogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Beane Freeman, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Research Triangle Institute, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Alavanja MC, Blair A, Merkle S, Teske J, Eaton B. Mortality among agricultural extension agents. Am J Ind Med. 1988;14(2):167-76. doi: 10.1002/ajim.4700140207. PMID 3207102
- [Background] Barthel E. Increased risk of lung cancer in pesticide-exposed male agricultural workers. J Toxicol Environ Health. 1981 Nov-Dec;8(5-6):1027-40. doi: 10.1080/15287398109530135. PMID 7338938
- [Background] Bjeldanes LF, Morris MM, Timourian H, Hatch FT. Effects of meat composition and cooking conditions on mutagen formation in fried ground beef. J Agric Food Chem. 1983 Jan-Feb;31(1):18-21. doi: 10.1021/jf00115a005. No abstract available. PMID 6826915
- [Derived] Lebov JF, Engel LS, Richardson D, Hogan SL, Hoppin JA, Sandler DP. Pesticide use and risk of end-stage renal disease among licensed pesticide applicators in the Agricultural Health Study. Occup Environ Med. 2016 Jan;73(1):3-12. doi: 10.1136/oemed-2014-102615. Epub 2015 Jul 15. PMID 26177651